CLINICAL TRIAL: NCT01613092
Title: Prevention of Arrhythmia Device Infection Trial (PADIT) Cluster Crossover Pilot Study
Brief Title: Prevention of Arrhythmia Device Infection Trial (PADIT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PADIT Cluster Crossover Pilot
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Arrhythmia
Keywords: Arrhythmia; Device Procedure; High risk patients; Antibiotics; Infection; Cluster
MeSH Terms: conditions — Arrhythmias, Cardiac; Infections | interventions — Cefazolin; Vancomycin; Bacitracin; Cephalexin; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Experimental): Preoperative Antibiotics
  Interventions: Drug: Cefazolin
- Aggressive (Incremental) (Active Comparator): Preoperative antibiotics, antibiotic wash and post operative antibiotics
  Interventions: Drug: Incremental

INTERVENTIONS:
Drug: Incremental — Cefazolin and Vancomycin pre-op, bacitracin wash and postoperative cefalexin or clindamycin
  Other Names: Cefazolin , Vancomycin, bacitracin, cefalexin or clindamycin
  Arms: Aggressive (Incremental)
Drug: Cefazolin — Preoperative antibiotic
  Arms: Conventional

SUMMARY:
The goal of the pilot study is to compare whether a centre-wide policy of incremental antibiotic therapy will reduce pacemaker infection compared to a policy of conventional antibiotic prophylaxis in high-risk patients undergoing arrhythmia device procedures. This pilot study will provide feasibility information for a larger cluster randomized crossover design (CRCD).

DETAILED DESCRIPTION:
Multi-center, cluster crossover, unblinded, pilot study. Centers will be randomized to conventional vs. incremental antibiotic therapy for 2 months or until eligible 20 patients are treated, whichever comes first. At 2 months, centers will have a crossover period of 4 weeks where the alternate strategy is implemented, followed by the final 2-month/20 patient enrolment period. During each treatment period the randomized antibiotic strategy will be used on all center patients undergoing a device implant procedure. Prior to the planned surgery or at the first follow up visit, patients who meet the study eligibility criteria will be approached to obtain consent for data collection purposes. Follow up will be according to usual clinical care at the center.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* received one of the following procedures:

  1. a second or subsequent procedure on the arrhythmia device pocket: i. ICD, pacemaker, CRT-P, CRT-D generator and/or lead replacement. ii. pocket or lead revision iii. system upgrade (insertion or attempted insertion of leads)
  2. new cardiac resynchronization therapy device implant (pacemaker or ICD)

Exclusion Criteria:

* life expectancy < 12 months in the opinion of the local investigator.
* allergy or unable to tolerate cefazolin or clindamycin or vancomycin.
* allergy or unable to tolerate intracavitary bacitracin identified per-operatively.
* pre-operative identification that the patient has infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hospitalization attributed to device infection | within one year of device procedure
  Hospitalization attributed to device infection

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Andrew Krahn, M.D, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Hamilton General Hospital, McMaster University, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario